CLINICAL TRIAL: NCT06830876
Title: Detecting Change in Muscle Parameters, Pain, and Function With Neuromuscular Electrical Stimulation Treatment in Individuals Living With Transtibial Amputation
Brief Title: Detecting Change in Muscle Parameters, Pain, and Function With NMES for TTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Peterson-Snyder (Industry)
Responsible Party: Sponsor-Investigator, Sara Peterson-Snyder, co-investigator, O&P Clinical Innovations
Organization: O&P Clinical Innovations (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMES-PIT-24
Record Dates: First submitted 2024-12-09; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-12

CONDITIONS: Amputation
Keywords: residual limb; pain; gait
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot study, with a one-group, repeated measures experiment with individuals with unilateral transtibial limb loss (n=20) who are independent ambulators. A repeated measures design is chosen to gather additional data efficiently, using the unaffected side as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NMES (Other): All participants will undergo an 8-week Neuromuscular Electrical Stimulation (NMES) intervention using a portable NMES device at home. Participants will use the device on their residual limb to stimulate specific muscle groups (vastus medialis oblique, tibialis anterior, and gastrocnemius muscles). Electrode placement, stimulation intensity, and session frequency will be standardized and tailored to each participant to achieve strong but tolerable muscle contractions.
  Interventions: Device: Chattanooga Continuum Device

INTERVENTIONS:
Device: Chattanooga Continuum Device — The Chattanooga Continuum (Enovis, Wilmington, DE) is an FDA-approved, multi-functional, dual-channel electrotherapy device that offers adjunctive rehabilitation therapies, including muscle re-education (NMES), pain control, and stimulation of local blood circulation. The device provides a treatment duration of up to 60 minutes, allowing for cycled or continuous therapy. It offers symmetrical and asymmetrical waveform types, adjustable pulse rates of up to 150 Hz, and pulse width durations of up to 400 μs. The device also features off times, channel ramp times, and on time settings. Additionally, the Continuum is equipped with a data and parameter logger, enabling the monitoring of patient usage. It incorporates an automatic lock function to prevent accidental changes in intensity by preventing unintended pressing of the control buttons. The device operates on two AA rechargeable NiMH batteries, and a battery charger and extra batteries are included with the device.
  Other Names: Continuum Device (EMPI)

SUMMARY:
The proposal aims to investigate a non-invasive, cost-effective method for rebuilding muscle mass in individuals with transtibial limb loss. Maintaining a healthy, pain-free residual limb is a primary concern for prosthesis users.

Amputees commonly experience muscle deficits leading to mobility issues, poor prosthetic fit, and chronic pain. Neuromuscular electrical stimulation (NMES) is a potential intervention that activates muscles with low-level electrical stimulation, improving strength, function, and reducing pain. The study seeks to understand NMES's effects on muscle parameters and pain to develop evidence-based interventions for amputees.

Twenty participants with transtibial amputations will undergo an 8-week NMES training program. Ultrasound imaging will assess muscle thickness, cross-sectional area, and composition changes. The study aims to enhance mobility, prosthetic fit, and overall well-being of amputees, addressing challenges and reducing healthcare burdens.

DETAILED DESCRIPTION:
This study investigates the efficacy of a home-based Neuromuscular Electrical Stimulation (NMES) intervention in improving muscle parameters, reducing pain, and enhancing gait biomechanics in individuals with unilateral transtibial amputation (TTA). Muscle atrophy and sarcopenia, common in individuals with amputations, result in reduced muscle strength, volume, and functional impairments. The NMES intervention aims to counter these deficits by promoting muscle hypertrophy and improving residual limb muscle quality.

Ultrasound (US) imaging, a safe and non-invasive technique, will be used to assess muscle composition and quality, focusing on muscle thickness (MT), cross-sectional area (CSA), and muscle fat infiltration (MFI) of key muscle groups, including the vastus medialis oblique (VMO), tibialis anterior (TA), and gastrocnemius (GM) muscles. Baseline measures will be compared to post-NMES intervention data to evaluate changes in muscle parameters.

Participants will undergo an 8-week NMES program using a portable device. Electrode placement and settings will be customized to target specific muscle groups for optimal stimulation and contraction. Anthropometric measurements, gait analysis, and self-reported pain levels will be collected at baseline, midpoint, and post-intervention. The study will utilize US imaging to validate changes in muscle composition and quality and examine improvements in gait parameters such as stride length, velocity, and step symmetry using the GAITRite® system.

This project is a critical step in addressing the lack of standardized rehabilitation protocols for individuals with TTA. By leveraging NMES and US imaging, the study aims to develop a cost-effective, accessible intervention that enhances prosthetic fit, stabilizes limb volume, and improves mobility. The findings will contribute to refining rehabilitation strategies and improving the quality of life for individuals with limb loss.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have a unilateral transtibial amputation
* Have normal sound limb range of motion and function
* Have a minimum of 4" length limb from tibial tubercle to end of residuum to allow room for NMES pads
* Report current pain at a level 3 or higher on a Visual Analog Scale (VAS)
* Pass a monofilament test on the residual limb in 7 out of 10 areas to ensure adequate sensation for NMES stimulation
* Have a body mass index (BMI) of 35 kg/cm2 or less as NMES works more effectively on lower BMI

Exclusion Criteria:

* Have used electrical stimulation on the residual limb in the past six months
* Have been diagnosed as a severe diabetic or self-report insensate skin
* Have the presence of open wounds/ulcers on the residual limb
* Have experienced a cerebrovascular accident (stroke) or nerve injury to a lower limb
* Wear a pacemaker or implanted cardiac defibrillator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine changes in muscle thickness changes via US imaging in the residual limb of the VMO, TA, and GM muscles after 8 -weeks of NMES at-home intervention | 9 months
  Compared to baseline, amputees' residual limb will show changes in Muscle Thickness (MT) measured in centimeters (cm) of the vastus medialis oblique (VMO), Tibialis Anterior (TA) and gastrocnemius muscles (GM) post-NMES intervention.

SECONDARY OUTCOMES:
To determine changes in muscle cross-sectional area (CSA) via US imaging in the residual limb of the VMO, TA, and GM muscles after 8 -weeks of NMES at-home intervention | 9 months
  Compared to baseline, amputees' residual limb will show changes in Muscle Cross-sectional area (CSA) measured in centimeters (cm) post-NMES intervention.
To determine changes in Muscle Fat Infiltration (MFI) or myosteatosis via US imaging in the residual limb of the VMO, TA, and GM muscles after 8 -weeks of NMES at-home intervention | 9 months
  Compared to baseline, amputees' residual limb will show changes in Muscle Fat Infiltration (MFI) or myosteatosis post-NMES intervention using values between 0 and 255 (0: black; 255: white) and scored with the Modified Heckmatt scale as z-scores.
To determine changes in chronic residual limb pain after 8 weeks of NMES at-home intervention. | 9 months
  NMES intervention will show changes in chronic residual limb pain after (post) intervention when compared to baseline (pre) as measured by a pain questionnaire designed for amputees measured using a numeric rating scale 0-10, 0 being no pain and 10 being the highest pain imaginable.
To determine changes in phantom limb pain after 8 weeks of NMES at-home intervention. | 9 months
  NMES intervention will show changes in phantom limb pain after (post) intervention when compared to baseline (pre) as measured by a pain questionnaire designed for amputees measured using a numeric rating scale 0-10, 0 being no pain and 10 being the highest pain imaginable.
To determine changes in phantom sensation after 8 weeks of NMES at-home intervention. | 9 months
  NMES intervention will show changes in phantom sensation after (post) intervention when compared to baseline (pre) as measured by a pain questionnaire designed for amputees measured using a numeric rating scale 0-10, 0 being no pain and 10 being the highest pain imaginable.
To determine changes in gait parameters of step length after (post) NMES at-home intervention when compared to baseline (pre) measures. | 9 months
  NMES intervention will show changes in gait parameters of step length in meters (post) intervention when compared to baseline (pre) measures with the use of a Gait Rite mat.
To determine changes in gait parameters in step width after (post) NMES at-home intervention when compared to baseline (pre) measures. | 9 months
  NMES intervention will show changes in gait parameters of step width in meters of the amputated side (post) intervention when compared to baseline (pre) measures with the use of a Gait Rite mat.
To determine changes in gait velocity after (post) NMES at-home intervention when compared to baseline (pre) measures. | 9 months
  NMES intervention will show changes in gait velocity (meters/time) after (post) intervention when compared to baseline (pre) measures with the use of a Gait Rite mat.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Leister, PhD, Principal Investigator — East Tennessee Sate University
Locations (1):
- Cranberry Township Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Snyder-Mackler L, Ladin Z, Schepsis AA, Young JC. Electrical stimulation of the thigh muscles after reconstruction of the anterior cruciate ligament. Effects of electrically elicited contraction of the quadriceps femoris and hamstring muscles on gait and on strength of the thigh muscles. J Bone Joint Surg Am. 1991 Aug;73(7):1025-36. PMID 1874764
- [Background] Talbot LA, Gaines JM, Ling SM, Metter EJ. A home-based protocol of electrical muscle stimulation for quadriceps muscle strength in older adults with osteoarthritis of the knee. J Rheumatol. 2003 Jul;30(7):1571-8. PMID 12858461